CLINICAL TRIAL: NCT06161636
Title: Contribution of the Kinematic Theory in the Early Differential Diagnosis of the Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Optina Diagnostics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 18.259
Record Dates: First submitted 2023-10-13; First posted 2023-12-08 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; Healthy; Parkinsonian Syndromes
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Parkinson Disease (PD): Participants will then have to perform three blocks of tests: the first focused on the scripted motor signature, a second on the voice signature, and a complementary block aimed at capturing the motor signature using gestures of greater amplitude.
  All the tests were designed to allow the characterization of the motor signature according to different aspects of motor control, but also to reproduce the same concepts in the three fields (scripted signature, voice signature and large amplitude motor signature), while allowing an acquisition of an approximate total duration of 30 minutes.
  For retinal photos, the subject's pupils will be dilated using eye drops (1% tropicamide and 2.5% phenylephrine) 15-20 minutes before taking the measurement. These drugs are considered the standard used by optometrists and ophthalmologists during pupil dilation.
- Patients with atypical Parkinsonian Syndromes (PS): Participants will then have to perform three blocks of tests: the first focused on the scripted motor signature, a second on the voice signature, and a complementary block aimed at capturing the motor signature using gestures of greater amplitude.
  All the tests were designed to allow the characterization of the motor signature according to different aspects of motor control, but also to reproduce the same concepts in the three fields (scripted signature, voice signature and large amplitude motor signature), while allowing an acquisition of an approximate total duration of 30 minutes.
  For retinal photos, the subject's pupils will be dilated using eye drops (1% tropicamide and 2.5% phenylephrine) 15-20 minutes before taking the measurement. These drugs are considered the standard used by optometrists and ophthalmologists during pupil dilation.
- Healthy volunteers: Participants will then have to perform three blocks of tests: the first focused on the scripted motor signature, a second on the voice signature, and a complementary block aimed at capturing the motor signature using gestures of greater amplitude.
  All the tests were designed to allow the characterization of the motor signature according to different aspects of motor control, but also to reproduce the same concepts in the three fields (scripted signature, voice signature and large amplitude motor signature), while allowing an acquisition of an approximate total duration of 30 minutes.
  For retinal photos, the subject's pupils will be dilated using eye drops (1% tropicamide and 2.5% phenylephrine) 15-20 minutes before taking the measurement. These drugs are considered the standard used by optometrists and ophthalmologists during pupil dilation.

SUMMARY:
The working hypotheses are as follows: #1 The processing of performance signals by automated lognormal segmentation and the extraction of the parameters of interest will make it possible to distinguish groups of patients from healthy elderly subjects. #2 The three instrumental approaches will not have the same degree of reliability as a predictive biomarker of clinical diagnosis established by consensus.

DETAILED DESCRIPTION:
The strength of this study is to compares three refined parametric approaches drawn from functions mediated by very different neuromuscular programs (visually guided voluntary movement control to perform trajectories with the hand or arm versus vocal control) among two groups of patients and a healthy group. Its weakness lies in the lack of multimodal methods to accurately confirm clinical diagnosis and the predictive reliability of patient performance. These modalities are too costly to be included in this project. However, different oculovisual measurement standards such as optical coherence tomography, hyperspectral imaging (OPTINA Diagnostics Inc.), and eye tracking will be used at the School of Optometry, University of Montreal. There is indeed a remodeling of the retina and oculomotor changes in Parkinson's Disease (PD) and these non-invasive techniques, which have been accepted for several years, will be used in patients in support of their clinical diagnosis compared to normal subjects.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Parkinsonism including idiopathic Parkinson's disease or a related syndrome;
* Have motor symptoms of Parkinsonism for 6 years or less;
* Be a healthy volunteer subject in good general health with no prior neurological history;
* Age between 50-75 years old;
* If applicable, be able to safely leave home in the morning without having taken antiparkinsonian medication for the past 12 hours.

Exclusion Criteria:

* Major neurocognitive disorders;
* History of other neurological conditions, such as ischemic or hemorrhagic stroke, paralysis of a limb, traumatic brain injury, epilepsy, orofacial dystonia, essential tremor;
* History of oromandibular or laryngeal procedures;
* Uncorrected deafness;
* Any contraindication to pupillary dilation.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sixty patients with Parkinson's disease (PD; N=30) or atypical Parkinsonian Syndromes (PS; N=30) will be recruited within the first 6 years of the disease. They will be recruited at the CHUM or from the Quebec Parkinson Network, and compared to healthy volunteers of comparable age (N=30). The atypical PS group will include people with multiple system atrophy or progressive supranuclear palsy. The probable final diagnosis of the two groups of patients will be confirmed by telephone contact two years after the research visit.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Lognormal primitives | Day 1
  Velocity profiles generated for simple movements (strokes) and certain vocal frequencies (formants), transformed to fit into the lognormal model

SECONDARY OUTCOMES:
Optical Coherence Tomography measures | Day 1
  Measures of thickness for macula, fovea, peripapillary retinal nerve fiber layer, divided in quadrants, expressed in microns.
Movement Disorder Society-Unified Parkinson's Disease Rating Scale section III | Day 1
  Motor rating in the practically defined unmedicated state, in points
Radboud Oral Motor Inventory for Parkinson's Disease | Day 1
  Clinical tool to evaluate perceived problems with speech, swallowing, and saliva in subjects with parkinsonism, in points

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Blanchet, Principal Investigator — CHUM/Université de Montréal
Locations (1):
- CHUM/Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spund B, Ding Y, Liu T, Selesnick I, Glazman S, Shrier EM, Bodis-Wollner I. Remodeling of the fovea in Parkinson disease. J Neural Transm (Vienna). 2013 May;120(5):745-53. doi: 10.1007/s00702-012-0909-5. Epub 2012 Dec 23. PMID 23263598
- [Background] Jimenez B, Ascaso FJ, Cristobal JA, Lopez del Val J. Development of a prediction formula of Parkinson disease severity by optical coherence tomography. Mov Disord. 2014 Jan;29(1):68-74. doi: 10.1002/mds.25747. Epub 2013 Nov 14. PMID 24458320